CLINICAL TRIAL: NCT07030959
Title: A Phase I Open-label, Multicenter Study to Evaluate the Safety, Pharmacokinetics, and Activity of AUBE00 in Patients With Solid Tumors
Brief Title: Study of AUBE00 in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AUB101CT
Record Dates: First submitted 2025-05-11; First posted 2025-06-22 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Dose Escalation part (Experimental): Patients will receive AUBE00 as an oral administration at escalated doses.
  Interventions: Drug: AUBE00
- Part B: Expansion part (Experimental): Patients will receive AUBE00 as an oral administration at multiple dose levels determined to be safe (including MTD).
  Interventions: Drug: AUBE00

INTERVENTIONS:
Drug: AUBE00 — AUBE00 as an oral administration

SUMMARY:
This is a first-in-human, Phase I, open-label, multicenter, multinational study, designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), immunogenicity, and anti-tumor activity of AUBE00 in patients with locally advanced or metastatic solid tumors.The total number of patients in this study will be approximately 70 to 100.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of signing Informed Consent Form (ICF)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients with Kirsten rat sarcoma (KRAS) alteration confirmed by local tests or central laboratory test (Details are defined for each part)
* Refractory or resistant to standard therapies or standard therapies are not available

Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant or breastfeeding during the study or within 27 weeks after the last dose of AUBE00
* Primary central nervous system (CNS) malignancy, untreated CNS metastases requiring any anti-tumor treatment, or active CNS metastases (progressing or requiring corticosteroids for symptomatic control)
* Significant cardiovascular disease, such as New York Heart Association (NYHA) Class II or greater cardiac disease, unstable angina, or myocardial infraction within the previous 6 months or unstable arrhythmias within the previous 3 months
* Patient with complications from a cerebrovascular disorder (such as subarachnoid hemorrhage, cerebral infarction, transient ischemic attack, etc.) or a history of such complications within 6 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events of AUBE00 [Part A, B] | From screening until study completion, treatment discontinuation or post-treatment follow up (up to approximately 49 months)
  Incidence, nature, and severity of adverse events (AEs), with severity determined according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0)
Number of participants with changes in vital signs of AUBE00 [Part A, B] | From screening until study completion, treatment discontinuation or post-treatment follow up (up to approximately 49 months)
  Change from baseline in vital signs (Includes respiratory rate, pulse oximetry, pulse rate, and systolic and diastolic blood pressure while the patient is in a seated or semi-recumbent position, and temperature.)
Number of participants with changes in clinical laboratory test of AUBE00 [Part A, B] | From screening until study completion, treatment discontinuation or post-treatment follow up (up to approximately 49 months)
  Change from baseline in clinical laboratory test
Number of participants with changes in Electrocardiograms (ECGs) of AUBE00 [Part A, B] | From screening until study completion, treatment discontinuation or post-treatment follow up (up to approximately 49 months)
  Change from baseline in ECGs (QT interval)
Maximum tolerated dose (MTD) of AUBE00 [Part A] | From Cycle 0 Day 1 until Cycle 2 Day 1 (approximately 30 days) (Cycle 0: 6 to 9 days, Cycle 1 and beyond each Cycle: 21 days)
  Incidence and nature of dose-limiting toxicities (DLTs)
Time to reach maximum plasma concentration (Tmax) of AUBE00 [Part A] | From Cycle 0 Day 1 until study completion, treatment discontinuation (up to approximately 49 months) (Cycle 0: 6 to 9 days, Cycle 1 and beyond each Cycle: 21 days)
  Tmax of AUBE00
Maximum plasma concentration (Cmax) of AUBE00 [Part A] | From Cycle 0 Day 1 until study completion, treatment discontinuation (up to approximately 49 months) (Cycle 0: 6 to 9 days, Cycle 1 and beyond each Cycle: 21 days)
  Cmax of AUBE00
Elimination half-life (t1/2) of AUBE00 [Part A] | From Cycle 0 Day 1 until study completion, treatment discontinuation (up to approximately 49 months) (Cycle 0: 6 to 9 days, Cycle 1 and beyond each Cycle: 21 days)
  t1/2 of AUBE00
Area under the plasma concentration-time curve (AUC) of AUBE00 [Part A] | From Cycle 0 Day 1 until study completion, treatment discontinuation (up to approximately 49 months) (Cycle 0: 6 to 9 days, Cycle 1 and beyond each Cycle: 21 days)
  AUC of AUBE00
Objective response of AUBE00 [Part B] | From screening until study completion, treatment discontinuation or post-treatment follow up (up to approximately 49 months)
  Objective response, defined as a confirmed complete response (CR) or partial response (PR) as the best overall response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as determined by the Investigator

SECONDARY OUTCOMES:
Objective response of AUBE00 [Part A] | From screening until study completion, treatment discontinuation or post-treatment follow up (up to approximately 49 months)
  Objective response, defined as a confirmed CR or PR as the best overall response per RECIST v1.1 as determined by the Investigator
Disease control of AUBE00 [Part A, B] | From screening until study completion, treatment discontinuation or post-treatment follow up (up to approximately 49 months)
  Disease control, defined as a confirmed CR, PR, or stable disease (SD) per RECIST v1.1 as determined by the Investigator
Duration of response (DoR) of AUBE00 [Part A, B] | From screening until study completion, treatment discontinuation or post-treatment follow up (up to approximately 49 months)
  DoR, defined as the time from the first occurrence of a documented objective response to the time of the first documented disease progression per RECIST v1.1 as determined by the Investigator or death due to any cause, whichever occurs first
Progression free survival (PFS) of AUBE00 [Part A, B] | From screening until study completion, treatment discontinuation or post-treatment follow up (up to approximately 49 months)
  PFS, defined as the time from the first study treatment to the first occurrence of disease progression per RECIST v1.1 as determined by the Investigator or death due to any cause, whichever occurs first
Anti-AUBE00 antibodies of AUBE00 [Part A, B] | From screening until study completion, treatment discontinuation or post-treatment follow up (up to approximately 49 months)
  Incidence of anti-AUBE00 antibodies
Overall survival (OS) of AUBE00 [Part B] | From screening until study completion, treatment discontinuation or post-treatment follow up (up to approximately 49 months)
  OS, defined as the time from the date of first study treatment to death due to any cause
Time to reach maximum plasma concentration (Tmax) of AUBE00 [Part B] | From Cycle 1 Day 1 until study completion, treatment discontinuation (up to approximately 49 months) (Cycle 1 and beyond each Cycle: 21 days)
  Tmax of AUBE00
Maximum plasma concentration (Cmax) of AUBE00 [Part B] | From Cycle 1 Day 1 until study completion, treatment discontinuation (up to approximately 49 months) (Cycle 1 and beyond each Cycle: 21 days)
  Cmax of AUBE00
Elimination half-life (t1/2) of AUBE00 [Part B] | From Cycle 1 Day 1 until study completion, treatment discontinuation (up to approximately 49 months) (Cycle 1 and beyond each Cycle: 21 days)
  t1/2 of AUBE00
Area under the plasma concentration-time curve (AUC) of AUBE00 [Part B] | From Cycle 1 Day 1 until study completion, treatment discontinuation (up to approximately 49 months) (Cycle 1 and beyond each Cycle: 21 days)
  AUC of AUBE00

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Chugai Pharmaceutical Co.Ltd, Study Director — clinical-trials@chugai-pharm.co.jp
Locations (4):
- United States (2):
  - South Texas Accelerated Research Therapeutics (START) Midwest, Grand Rapids, Michigan
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform. For further details on Chugai's Data Sharing Policy and how to request access to related clinical study documents, see here (www.chugai-pharm.co.jp/english/profile/rd/ctds_request.html).